CLINICAL TRIAL: NCT06458400
Title: To Evaluate the Efficacy and Safety of Tegileridine and Oliceridine Injections in the Treatment of Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuwei Qiu (Other)
Responsible Party: Sponsor-Investigator, Yuwei Qiu, Associate chief physician, Associate director of anesthesiology, Associate professor, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGRD-ANAL-PILOT-001
Record Dates: First submitted 2024-05-26; First posted 2024-06-13 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Analgesia
Keywords: Analgesia; Biased μ-opioid receptor agonists
MeSH Terms: conditions — Agnosia | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tegileridine (Experimental): The loading iv dose: 0.75mg The PCIA dose：0.05mg Lockout time: 10min
  Interventions: Drug: Tegileridine
- oliceridine (Experimental): The loading iv dose: 1.5mg The PCIA dose：0.35mg Lockout time: 6min
  Interventions: Drug: Oliceridine
- morphine (Active Comparator): The loading iv dose: 3mg The PCIA dose：1mg Lockout time: 6min
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Tegileridine — single dose+PCA dose
  Arms: tegileridine
Drug: Oliceridine — single dose+PCA dose
  Arms: oliceridine
Drug: Morphine — single dose+PCA dose
  Arms: morphine

SUMMARY:
This was a single-center, randomized, open-label, controlled exploratory study conducted in Chinese patients. The study planned to enroll Chinese patients to evaluate the efficacy and safety of tegileridine and oliceridine injection in the treatment of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Accept elective laparoscopic combined thoracic surgery under general anesthesia, surgery time ≥ 1 h;
2. 18 years old ≤ age ≤70 years old, regardless of gender;
3. 18 kg/m2≤BMI≤30 kg/m2;
4. American Society of Anesthesiologists (ASA) grade ⅰ-ⅲ;
5. Within 4 hours after the end of surgery, NRS≥4 in the resting state at any time;
6. Before starting trial-related activities, participants should voluntarily sign the informed consent form, fully understand the purpose and significance of this trial, and voluntarily abide by the trial procedures.

Exclusion Criteria:

1. Patients with a previous history of difficult airway (obstructive sleep apnea syndrome), severe respiratory depression such as oxygen saturation < 90%, or a history of acute or severe bronchial asthma;
2. Patients with a history of severe cardiovascular and cerebrovascular diseases (such as myocardial infarction or unstable angina pectoris, or severe arrhythmia such as atrioventricular block of degree Ⅱ or above, or ischemic stroke in NYHA class Ⅱ or above);
3. Known or suspected gastric bowel obstruction, including paralytic ileus patients;
4. Patients with allergy to opioids or any component of the trial drug;
5. Subjects with previous psychiatric disorders (such as schizophrenia, depression, etc.) and cognitive impairment;
6. With late-stage malignant tumors or with extensive metastasis of malignant tumor patients;
7. Subjects with other somatic pain that may affect postoperative pain assessment;
8. A history of drug, drug, and/or alcohol abuse within 1 year before randomization;
9. Pregnant or lactating female subjects;
10. Subjects with any other factor considered by the investigator to be ineligible for participation in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Time-weighted sum of differences of resting pain score within 24 hours after starting a loading dose of test drug infusion | during the first 24 hours after starting a loading dose of test drug infusion
  "resting pain score" is assessed by Numeric Rating Scale, range 0-10, 0=no pain and 10 = worst imaginable pain, from 0 to 0 means worse pain

SECONDARY OUTCOMES:
Resting-state pain and exercise-state pain intensity | Pain scores are evaluated at 10 minutes、30 minutes、6 hours、12 hours、24 hours after the first loading dose
  Resting-state pain and exercise-state pain intensity are assessed by Numeric Rating Scale, range 0-10, 0=no pain and 10 = worst imaginable pain, from 0 to 0 means worse pain
Time-weighted sum of differences of exercise-state pain score within 24 hours after starting a loading dose of test drug infusion | Pain scores are evaluated at 10 minutes、30 minutes、6 hours、12 hours、24 hours after the first loading dose
  "exercise-state pain score" is assessed by Numeric Rating Scale, range 0-10, 0=no pain and
total pain relief (TOTPAR) scores | 10 minutes、30 minutes、6 hours、12 hours、24 hours after the first loading dose
  Time-weighted sum of resting and moving state pain relief scores
the percentage of patients receiving rescue analgesia | from 0-24 hours after the first loading dose
  the percentage of patients receiving rescue analgesia
length of bed stay | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 1 months.
  length out of bed
Length of hospital stay | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 1 months.
  postoperative length of hospital stay
incidence of Postoperative nausea and vomiting | the first 24 hours after surgery
  incidence rate of PONV
incidence rate of respiratory depression | the first 24 hours after surgery
  respiratory depression is defined as respiratory rate < 8 and/or SpO2<90%
analgesia satisfaction | the first 24 hours after surgery
  satisfaction evaluation using 0-100 scale
pressing times of postoperative analgesic pump | the first 24 hours after surgery
total doses of postoperative analgesic pump | the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- 241 Huaihai West Road, Xuhui District, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Share when necessary